CLINICAL TRIAL: NCT06696118
Title: Electromagnetic Transduction Therapy (EMTT) on Mid-foot Osteoarthritis: A Pilot Study
Brief Title: Electromagnetic Transduction Therapy on Osteoarthritis in the Foot and Ankle
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Elizabeth Bondi, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-002661
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-07

CONDITIONS: Osteoarthritis Ankle; Osteoarthritis Foot
Keywords: Electromagnetic Transduction Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Mid-foot osteoarthritis (Experimental)
  Interventions: Device: Electromagnetic Transduction Therapy (EMTT)

INTERVENTIONS:
Device: Electromagnetic Transduction Therapy (EMTT) — Subjects will be treated with Electromagnetic Transduction Therapy (EMTT) using the Curamedix MAGNETOLITH device. Treatments will be administered twice per week, for four weeks. Each treatment will have the following settings: level 8, 8Hz, and 10,000 pulses andwill take about 15 to 20 minutes. Treatments will be spaced 2-3 days apart.

SUMMARY:
The purpose of this study is to determine if Electromagnetic Transduction Therapy (EMTT) is a viable treatment option in patients with osteoarthritis of the foot and/or ankle.

ELIGIBILITY:
Inclusion Criteria:

• Men and women with osteoarthritis of the foot and/or ankle confirmed via radiographs.

Exclusion Criteria:

• Pacemaker, active cancer, shrapnel, metal in eye, implantable devices that are not compatible with MRIs, concurrent foot or ankle condition or injury, prior foot or ankle surgery for osteoarthritis, steroid, platelet rich plasma, or hyaluronic acid injection within 2 months of the treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03-13 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) for Pain | Baseline, 3 weeks, 3 months, 6 months
  The VAS is a 11-item questionnaire assessing pain. Using a scale of 0 = no pain to 10 = worst pain. Total scores range from 0 - 110, lower scores indicating lower pain and higher scores indicating greater pain.
Foot and Ankle Ability Measure (FAAM) | Baseline, 3 weeks, 3 months, 6 months
  The Foot and Ankle Ability Measure (FAAM) ADL is a 21-item self-report questionnaire measuring Activities of Daily Living. Each item is scored on a 5-point Likert scale (4 to 0) from 'no difficulty at all' to 'unable to do'. Item score totals, which range from 0 to 84 are reported in percentage scores. Higher scores represent higher levels of function, with 100% representing no dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Bondi, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No